CLINICAL TRIAL: NCT06514482
Title: Registro español de Pacientes Con Apnea Del sueño y Somnolencia Diurna
Brief Title: Spanish Registry of Patients With Sleep Apnea and Daytime Sleepiness
Acronym: HYPNOSA
Status: Recruiting | Type: Observational
Sponsor: Hospital San Pedro de Logroño (Other)
Responsible Party: Sponsor
Other Study IDs: PI 569
Record Dates: First submitted 2023-08-02; First posted 2024-07-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea
Keywords: CPAP, residual sleepiness, OSA
MeSH Terms: conditions — Sleep Apnea Syndromes; Microcephaly, Primary Autosomal Recessive, 6; Sleep Apnea, Obstructive | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- NO OSA: Control group
  Interventions: Diagnostic Test: Diagnosis
- OSA WHITH CPAP
  Interventions: Diagnostic Test: Diagnosis
- OSA WHITHOUT CPAP
  Interventions: Diagnostic Test: Diagnosis

INTERVENTIONS:
Diagnostic Test: Diagnosis — Diagnosis

SUMMARY:
Multicenter, observational and prospective study, in which patients referred to the sleep unit with suspected apnea will be recruited obstructive sleep. 1000 patients referred to the sleep unit will be recruited with suspected obstructive sleep apnea. The recruited patients will undergo a sleep study for the diagnosis of OSA, ambulatory monitoring of blood pressure (ABP) of 24 hours, clinical variables will be obtained, questionnaires of quality of life, Epworth test for the evaluation of daytime sleepiness, variables biochemistry and obtaining biological samples. OSA patients will be managed following the usual practice. In those patients for whom the treatment with CPAP an evaluation of adherence to treatment will be carried out.

OSA patients will be evaluated at baseline, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who come to the sleep consultation for sleep study results for suspected OSA.
* Patients older than 18 years.
* Signature of the informed consent.

Exclusion Criteria:

* Psycho-physical inability to complete questionnaires.
* Presence of any previously diagnosed sleep disorder: narcolepsy, insomnia, sleep deprivation (less than 6h/day), regular use of medications hypnotics or sedatives (may be included if you only use a short-acting benzodiazepine or melatonin) and restless legs syndrome.
* Patients with > 50% central apnea or presence of Cheyne-Stokes respiration (CSRsp).
* A medical history that may interfere with the objectives of the study or that in the judgment of the investigator compromises the conclusions.
* Any medical, social or geographical factor that may endanger the patient compliance. (eg, alcohol consumption (more than 80 g/day in men and more than 60 gr / day in women), absence of stable habitual residence, disorientation or non-compliance history).
* Any process, cardiovascular or not, that limits life expectancy to less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the sleep unit with suspected obstructive sleep apnea dream.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 6 months
  Data analysis of the AHI in the respiratory polygraphy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Pedro, Logroño, La Rioja, Spain

IPD SHARING:
Plan to Share IPD: Undecided